CLINICAL TRIAL: NCT04880928
Title: Prospective Intraindividual Comparison of the Mydriasis of a Standardized Intracameral Anaesthetics With the Topical Preoperative Drop Application in the Uncomplicated Cataract Surgery
Brief Title: Comparison Mydriasis by Mydrane With Topical Drop Application
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Mydriasis with Mydrane
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Injections, Intraocular; Ophthalmic Solutions; Tropicamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injection solution (Experimental): Mydrane, Tropicamid 0,02%, Phenylephrine 0,31%, Lidocain 1%, injection solution
  Interventions: Drug: Eye injection (Mydrane)
- Standard eye Drops (Active Comparator): Phenylephrine 10% and Tropicamid 0,5% eye drops
  Interventions: Drug: eye drops (Phenylephrin); Drug: eye drops (Tropicamid)

INTERVENTIONS:
Drug: Eye injection (Mydrane) — Mydrane 0.2 mg/ml + 3.1 mg/ml
  + 10 mg/ml solution for injection tropicamide / phenylephrine hydrochloride / lidocaine hydrochloride
  Other Names: Mydrane
  Arms: injection solution
Drug: eye drops (Phenylephrin) — Phenylephrine 10%
  Other Names: Minims
  Arms: Standard eye Drops
Drug: eye drops (Tropicamid) — Tropicamid 0,5%
  Other Names: Agepha
  Arms: Standard eye Drops

SUMMARY:
The primary aim of the study is to compare the effectiveness of the intracameral application of Mydrane® (standardized combination of Tropicamide 0.02%, Phenylephrine 0.31% and Lidocaine 1%) with the preoperative topical application (Tropicamide 0.5% and Phenylephrine 10%). To evaluate the steadiness of the dilating effect on the pupil, the ratio of eyes without necessity for further pupil dilating procedures to perform the capsulorhexis is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the age of 50 to 100 years
* Day-hospital and inpatient care
* Clinically significant opacity of the lens with indication for cataract surgery on both eyes
* Lack of previous ophthalmic surgeries
* Lack of relevant ophthalmic conditions: Pseudoexfoliation syndrome, eye injuries, present inflammation (in terms of uveitis, endophthalmitis and iridocyclitis), restricted mydriasis (pupil diameter below 7mm after application of tropicamide 0.38% and phenylephrine HCL 2.5% - at preoperative examination), elevated intraocular pressure, alpha-receptor inhibitor intake (e.g. tamsulosin) due to impeded mydriasis

Exclusion Criteria:

* Allergic to phenylephrine, tropicamide, sodium metabisulfite, disodium edetate, sodium hydroxide, hydrochloric acid, lidocaine hydrochloride, sodium chloride, disodium phosphate dodecahydrate, disodium phosphate dihydrate
* Allergic to anesthesia (amide type)
* Allergic to atropine derivates
* Heart disease, tachycardia, hypertensive crises
* Aneurism of big vessels
* Untreated hyperthyroidism
* Untreated closed angle glaucoma and narrow angles with tendencies to glaucoma by intake of mydriatic drugs
* Pregnancy, breast feeding and premenopausal women

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
pupil dilating | during first and second surgery: a maximum of four weeks between first and second surgery
  The frequency of the feasibility of capsulorhexis without additional pupil dilating actions

SECONDARY OUTCOMES:
subjective highest intraoperative pain | after first and second surgery: a maximum of four weeks between first and second surgery
  Highest intraoperative pain visualized on a visual analogue scale (VAS) asked by a questionnaire, with the minimum 1 and maximum 10 , where higher scores mean a worse outcome
subjective perception of anesthetic procedures | after first and second surgery: a maximum of four weeks between first and second surgery
  perception of anesthetic procedures visualized on a visual analogue scale (VAS) asked by a questionnaire, with the minimum 1 and maximum 10 , where higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No